CLINICAL TRIAL: NCT02795039
Title: Open-label, Two-treatment, Single Period, Parallel, Single-dose, Randomized, Fasting, Lab-blinded Bioequivalence Study of Fulvestrant 50 mg/mL Versus Faslodex®, 50 mg/mL, in Healthy, Post-menopausal Female Subjects
Brief Title: Bioequivalence Study of Fulvestrant Injection 50 mg/mL in Healthy Post-menopausal Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FULV-006-CP1
Record Dates: First submitted 2016-05-30; First posted 2016-06-09 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2016-07

CONDITIONS: Healthy
MeSH Terms: interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fulvestrant 50mg/mL (Fresenius Kabi) (Experimental): 5 mL intramuscular injection
  Interventions: Drug: Fulvestrant
- Fulvestrant 50 mg/mL (Faslodex®) (Active Comparator): 5 mL intramuscular injection
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — Single 5 mL intramuscular injection (slowly over 1-2 minutes) of Fulvestrant into the right buttock (upper outer quadrant)
  Arms: Fulvestrant 50mg/mL (Fresenius Kabi)
Drug: Fulvestrant — Single 5 mL intramuscular injection (slowly over 1-2 minutes) of Faslodex® (Fulvestrant) into the right buttock (upper outer quadrant)
  Other Names: Faslodex
  Arms: Fulvestrant 50 mg/mL (Faslodex®)

SUMMARY:
The purpose of this study is to demonstrate bioequivalence between the test drug product, fulvestrant Injection, 50 mg/mL, and the Reference Listed Drug, Faslodex® Injection, 50 mg/mL.

DETAILED DESCRIPTION:
This study is being conducted to establish bioequivalence between sponsor's test product [fulvestrant Injection, 50 mg/mL (Manufactured for Fresenius Kabi, USA)] and reference listed drug [Faslodex® Injection, 50 mg/mL, (Distributed by AstraZeneca Pharmaceuticals, USA] after intramuscular administration of a 250 mg dose (5 mL injection) into the upper outer quadrant of the right buttock to normal, healthy, nonsmoking post-menopausal female subjects.

The order of receiving the test product (T) or reference listed drug (R) for each subject during the study will be determined according to a randomization schedule.

Subjects will be allocated with a ratio of 1:1 to both treatment groups (i.e. T and R).

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy, non smoking post-menopausal female subjects between the ages of 40 and 65 years (inclusive) Note: Postmenopausal is defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL. The amenorrhea should not be due to lactation
* Body Mass Index (BMI = weight/height2) greater than or equal to 18.5 kg/m2 and less than or equal to 29.9 kg/m2
* Physical examination, 12-lead electrocardiogram (ECG) and vital signs without any clinically significant findings
* Negative for urine drugs of abuse screen, urine nicotine (cotinine) screen, and breath alcohol screen.
* Negative for hepatitis B-surface antigen, hepatitis C and Human Immunodeficiency Virus (HIV)
* Clinical laboratory values within the acceptable range, unless deemed clinically not significant by the principal investigator or sub-investigator.
* Availability of the subject for the entire study period and willingness of the subject to adhere to protocol requirements as evidenced by signing the Informed Consent Form (ICF).

Exclusion Criteria:

* History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, musculoskeletal, psychiatric, or cardiovascular disease or malignancies or any other condition which, in the opinion of the principal investigator or sub-investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* A history of allergic or adverse response(s) to fulvestrant, castor oil, benzyl alcohol, benzyl benzoate, polysorbate 80, α-tocopherol or any other comparable or similar products.
* Smoking or use of tobacco products within 6 months prior to the first dose of study drug or during the study
* Positive urine pregnancy test at screening or serum pregnancy test prior to administration of study drug.
* History of any bleeding disorders
* Consumption of alcohol exceeding 10 drinks/ week in the previous 1 year
* Intolerance to/fear of venipuncture, needles or blood draws
* Have consumed any products or undergone any procedures mentioned under "restriction table" in protocol
* Surgically-induced post menopausal females

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration | 0-238 days
Area under the plasma concentration versus time curve (AUC0-238d) of fulvestrant | 0-238 days

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC0-28d) of fulvestrant | 0-28 day
Area under the plasma concentration versus time curve from time zero to the last measurable concentration (AUC0-t) | 0-238 days
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC0-∞) | 0-238 days
Time to Reach the Maximum Plasma Concentration (Tmax) | 0-238 days
Elimination Half-life Period (t1/2) | 0-238 days
Terminal Slope (λz) | 0-238 days
Residual area in percentage (AUC_%Extrap_obs) | 0-238 days
Injection site pain assessment | 0-8 days

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Lambda Therapeutic Research Inc., Toronto, Ontario
  - BioPharma Services Inc., Toronto, Ontario
  - Algorithme Pharma Inc., Mount Royal, Quebec

IPD SHARING:
Plan to Share IPD: No